CLINICAL TRIAL: NCT06918483
Title: An Evaluation of Care (Education) and Treatment Reviews for People With Learning Disabilities and Autistic People (CECILIA)
Brief Title: An Evaluation of Care (Education) and Treatment Reviews for People With Learning Disabilities and Autistic People
Acronym: CECiLiA
Status: Not yet recruiting | Type: Observational
Sponsor: Coventry and Warwickshire Partnership NHS Trust (Other Government)
Collaborators: University of Birmingham (Other); University of East Anglia (Other); University of Kent (Other); Learning Disability England (Unknown); The National Autistic Society (Unknown); The Challenging Behaviour Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 350098; NIHR 158265 (Other Grant/Funding Number: National Institute for Health and Care Research: Health and Social Care Delivery Research (HSDR) programme)
Record Dates: First submitted 2025-04-01; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder; Intellectual Disabilities
Keywords: Care (Education) and treatment reviews (C(E)TRs); Autistic people; People with an intellectual disability
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 695 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- A person with a learning disability, or an autistic person: Inclusion criteria:
  A person with a learning disability, or an autistic person who has received or taken part in a C(E)TR within the last 12-months including Blue Light (community) C(E)TRs; is aged 5 or older (i.e. eligible to attend school at Key Stage one) For those aged 16 years and older who lack capacity to make a decision about taking part in this research, advice indicating that they should be included from either a personal or nominate consultee For those aged 15 and younger, consent from the person or organisation with parental responsibility
  Exclusion criteria:
  Only having received or taken part in Independently Chaired Care (Education) and Treatment Reviews (IC(E)TRs) within the last 12-months. IC(E)TRs are only for those held within long-term segregation and are out of scope Anyone aged younger than 5 years
- A family member or carer of an autistic person or person with a learning disability: Inclusion criteria:
  A family member or carer of an autistic person or person with a learning disability who has 1. received or taken part in a C(E)TR within the last 12-months including blue-light C(E)TRs and 2. is aged 5 or older (i.e. eligible to attend school at Key Stage one).
  Exclusion criteria:
  1. A family member or carer of an autistic person or person with a learning disability who has only having received or taken part in Independently Chaired Care (Education) and Treatment Reviews (IC(E)TRs) within the last 12-months. IC(E)TRs are only for those held within long-term segregation and are out of scope; or who is aged younger than 5 years.
- A C(E)TR panel member (Chair, Expert by Experience or clinical member): Inclusion criteria:
  A C(E)TR panel member who has taken part in a C(E)TR within the last 12-months including blue-light C(E)TRs.
  Exclusion criteria:
  Staff who have only taken part in Independently Chaired Care (Education) and Treatment Reviews (IC(E)TRs) within the last 12-months. IC(E)TRs are only for those held within long-term segregation and are out of scope
- Health and social care professional (including commissioners): Inclusion criteria:
  A health or social care professional, or commissioner who has taken part in a C(E)TR within the last 12-months including blue-light C(E)TRs.
  Exclusion criteria:
  Staff who have only taken part in Independently Chaired Care (Education) and Treatment Reviews (IC(E)TRs) within the last 12-months. IC(E)TRs are only for those held within long-term segregation and are out of scope

SUMMARY:
Aims In this research project, we will determine whether Care (Education) and Treatment Reviews are helpful for people with learning disabilities and autistic people and their families.

Background Care (Education) and Treatment Reviews were started in 2014 to help get autistic people and people with learning disabilities out of psychiatric hospitals and to prevent their admission to psychiatric hospitals. Care (Education) and Treatment Reviews involve an independent panel including an Expert by Experience, a clinician, and a commissioner who is responsible for paying for an individual's care. The autistic person or the person with learning disability and their family also attend the meeting. The focus of a Care (Education) and Treatment Review is to either prevent a person from being admitted to a psychiatric hospital in the first place, or to help someone who is already in hospital, get out. They do this by trying to work out ways to overcome barriers that might be stopping someone from leaving hospital. However, we do not know if Care (Education) and Treatment Reviews stop people from being admitted to a psychiatric hospital in the first place, or help people already in hospital get out.

Method Our project has four stages. In Stage 1 we will work with the members of our Lived Experience Advisory Panels to co-produce survey questions. We will design surveys for people with learning disabilities and autistic people, families and carers, Care (Education) and Treatment Reviews panel members, and health and social care professionals to complete. We will share these surveys with as many people as we can nationally. We will make adjustments so that people with learning disabilities can take part in our surveys. We know that individuals with moderate to severe learning disabilities and younger children will not be able to complete the surveys and so we will use other ways to gather their views and experiences. We will also try to work out how much it costs to have a Care (Education) and Treatment Review .

Within Stage 2, we will find out how patients in hospital are doing over time, by attending Care (Education) and Treatment Reviews, CPA, and other patient meetings. We will ask people, including people with moderate and severe learning disabilities to take part in some interviews with us, ensuring we adapt the interview process, so it is accessible. We will use the information from these interviews to work out whether Care (Education) and Treatment Reviews are helping people and making things better.

In Stage 3, we will look at the anonymous data that is collected by the NHS about everyone with a learning disability or autism who is admitted to hospital. We will work out what sorts of things helped them and what sorts of things did not help them get out of hospital. We think we will have data that covers over 11 years.

Within our final stage, Stage 4, we will bring together all of the information we have collected from the different stages of the research to work out what it tells us. We will use the information along with input from our Lived Experience Advisory Panel members to co-produce and share reports and information about what we have found out. We will also co- develop and publish good practice guidance for doing Care (Education) and Treatment Reviews and make sure our guidance is shared in different ways and to different people who need it.

Patient/public involvement We have partnered with Learning Disability England, the National Autistic Society, and the Challenging Behaviour Foundation who will each lead one of our three Lived Experience Advisory Panels: (1) people with learning disabilities, (2) autistic people, and (3) carers and family members. We will have regular meetings with each Lived Experience Advisory Panel to make sure we they can provide input throughout the study. They will help us to design the surveys and interviews, interpret our findings, share the findings and co-produce and publish our good practice guidance in different formats for different target audiences. Each advisory panel will meet separately but we will bring them together once a year to benefit from their combined input.

Our project has been developed collaboratively with Learning Disability England, the National Autistic Society, and the Challenging Behaviour Foundation who all have experience of being involved within Care (Education) and Treatment Reviews. Learning Disability England, the National Autistic Society, and the Challenging Behaviour Foundation will be core members of our study management and study steering committees. Further, a nurse with significant learning disability and autism experience, Expert-by-Experience, and Care (Education) and Treatment Review panel chair is a co-researcher. A carer of a man with severe learning disability is also a co-researcher.

DETAILED DESCRIPTION:
Aim To undertake an evaluation of C(E)TRs using mixed methods across four stages with five work packages with children and adults with learning disabilities and autistic children and adults across a range of inpatient settings, including those in the community who receive a C(E)TR who are at risk of admission

Objectives

1. To understand the experiences of all stakeholders, including people with learning disabilities and autistic people and their families, when taking part in C(E)TRs including descriptions of the barriers and facilitators to genuine participation and the use of augmentative and alternative communication, and options for improvement.
2. To understand how C(E)TRs are being carried out in practice with a range of people with learning disabilities and autistic people across different settings, including those at risk of admission who are in the community.
3. To understand how C(E)TRs may be changing care pathways, improving outcomes, potentially preventing admission or promoting discharge, their possible cost implications, and how this is different from existing methods for reviewing care, and to make recommendations for improvement.
4. To publish good practice guidance inclusive of practical resources and tools for conducting C(E)TRs and outcome implementation, including how to promote inclusion and participation for people with learning disabilities and autistic people

Research questions

1. What are the experiences of people with learning disabilities and autistic people, families, C(E)TR panel members and a range of health and social care professionals when taking part in C(E)TRs?
2. How are experts by experience being included and supported to take part in C(E)TRs? What are the barriers and facilitators to participation and how can their participation be promoted?
3. How are C(E)TRs being carried out in practice with different groups (e.g., children, adults, autistic adults without learning disabilities) and in different settings (e.g., assessment and treatment units, secure units, acute mental health wards, inpatient units for children)?
4. What impact do C(E)TRs have upon care-pathways, and how are recommendations and outcomes implemented and monitored?
5. What barriers and facilitators to discharge are identified by C(E)TRs and how are they overcome or addressed by care teams?
6. How are C(E)TRs different, similar to, or integrated with existing methods for reviewing care (e.g., Care Programme Approach, Child Protection Conferences, Extraordinary Care Review Meetings)?
7. How are C(E)TRs structured and managed to support inclusion, and what adjustments and supports aid participation (e.g., augmentative and alternative communication) of people with learning disabilities and autistic people, and how can these be improved?
8. Is there evidence that people with learning disabilities and autistic people who are receiving a C(E)TR are being empowered as a consequence of C(E)TRs? What are the barriers and facilitators to empowerment and how can this be promoted?
9. Is there a relationship between the skill mix of a C(E)TR panel and the recommendations or outcomes made and are they implemented and how?
10. Are C(E)TRs associated with reducing inpatient numbers and what effect do they have on costs?
11. What are likely resource implications of C(E)TR and how might they differ between different types of individuals?

    Study design This research has four stages comprising five work packages using mixed methods. Lived Experience Advisory Panels (LEAPs) will co-produce study materials and will be actively engaged throughout each stage and all work packages. Initially, the investigators will co-develop a logic model informed by existing guidance and other literature to describe C(E)TR key activities, mechanisms of change, and outcomes which will be used to inform the choice of survey and interview questions and analysis within Stages 1 and 2, the analytic strategy within Stage 3, and the data triangulation within Stage 4. A logic model will be developed in collaboration with Lived Experience Advisory Panels (LEAPs) and the Study Management Group inclusive of C(E)TR panel members. The investigators will also seek direct feedback from lead staff in NHS England who lead C(E)TR policy.

    Within Stage 1, national surveys) will be circulated to people with learning disabilities and autistic people, including children and young people, families and carers, C(E)TR panel members, and health and social care professionals. Surveys will ask about their experiences of taking part in C(E)TRs and also gather data to inform estimates of the likely cost of undertaking C(E)TRS. The investigators will use adapted methods, led by expert partners and with LEAP input to capture the voice of younger children and those with moderate-severe learning disabilities and those with associated communication difficulties including children and young people whose views and experiences are often not collected.

    Within Stage 2, the investigators will attend C(E)TRs, and CPA meetings to track individual progress over time, collect naturalistic data from the meetings, and undertake semi-structured interviews with attendees. The investigators will undertake a linguistic analysis of the data to determine the relative contributions of different individuals to the decision-making process, and the investigators will develop a descriptive temporal pathway model of C(E)TRs process over time and determine how C(E)TRs affect care pathways.

    In Stage 3, the investigators will model relationships between C(E)TRs and numbers of admissions, discharges, total number of inpatients, types of inpatient service, consider cost-implications and length of stay over time using anonymised data available from NHS Digital for children and adults.

    Within the final stage, Stage 4, the investigators will combine their quantitative and qualitative data to generate conclusions and develop and publish good practice guidance and practical resources and tools (e.g., videos, easy to read checklists, guides to promote good communication) for C(E)TRs including outlining best practice for maximising participation and engagement

    Participant selection Stage 1 (Work Package 1) The survey sample will include key sub-groups of the population of autistic people, people with learning disabilities, and their carers and family members. The investigators will ensure this by explicitly sampling younger and older autistic people and younger and older people with learning disabilities nationally who are receiving a service from a variety of services including inpatient and community services, forensic services, services for children and adolescents, acute and non-specialist services, and community learning disabilities teams. The investigators will capture data about protected characteristics including the nature and degree of disability, ethnicity, age, and sex, and if needed, revise the recruitment strategy to help ensure that the final sample includes participants from key sub-groups.

    Children aged 5 and above (eligible for entry to school Key Stage 1) will be included because evidence suggests rarely very young autistic children or children with learning disabilities are at risk of admission or are admitted to a specialist psychiatric hospital. The investigators anticipate that younger children will be unable to complete the survey and will make use of a highly structured approach to capture their voice when possible. The study needs to include the full range of individuals that may have experience of a C(E)TR, and will intentionally sample from ethnically diverse regions (e.g., urban areas with large diverse communities) to help ensure that the sample is suitable to examine associations with ethnicity. Study materials will be available in different languages and interviews can be completed with a translator.

    The investigators will make appropriate adaptations to meet the communication needs of people with learning disabilities or autistic people (e.g., easier-to-read text, pictorial prompts, having a supporter present, embedded text to speech reader, manual signing) including offering people the option of completing the survey together with a researcher either online or in person. The investigators will include a version for older children and young people which can be completed with additional support. It is likely the case that some older children and teenagers with mild learning disabilities will be able to complete an online version of the survey with limited support. However, this will likely not be the case for some, including younger children. For this group, who are not able to complete a survey, the option of completing a Talking Mats® interview will be offered instead. For those with no or limited vision, further adaptations will be made (e.g., visually enhanced rating scale with optional tactile markers for completion in person, and/or embedded text-to-speech functions for online completion).

    Running in parallel with the surveys, the investigators will complete structured interviews with a minimum of 25 people with learning disabilities and autistic people who have moderate to severe learning disabilities including children and adolescents with moderate to severe learning disabilities. These participants will be in addition to the minimum of 150 people with learning disabilities or autistic people who will complete the survey. Those with moderate to severe learning disabilities are likely unable to take part in the survey except through the participation of their carers. To capture their voice directly, the investigators will make use of augmentative and alternative communication methods to support the communication of participants as appropriate to their needs, such as Talking Mats® (www.talkingmats.com) and manual sign support (https://makaton.org). These participants are likely to lack capacity to make a decision about whether they wish to take part in the survey.

    Stage 1 (Work Package 2) The sample will include key sub-groups of the C(E)TR workforce and health and social care professionals. The study will recruit participants from both urban and rural areas within England across the full range of professionals who are involved in C(E)TRs. This includes paid and unpaid care staff along with professional staff and Experts by Experience (EbEs). Data about protected characteristics including disability, ethnicity, age, and sex will be captured. If needed, the recruitment strategy will be revised to ensure that the final sample contains sufficient data from key sub-groups. If required, materials will be translated and associated costs have been included. The investigators will provide participants with the option to complete the survey with a researcher, which may be helpful for EbEs, and will help ensure full participation.

    Stage 2 (Work Package 3) The study will recruit potential participants from across England within three broad regions: (a) eastern, (b) southeastern and southwestern, and (c) midlands and northern incorporating urban and rural locations across a range of inpatient services to ensure that the sample includes key sub-groups of the wider population of autistic people and people with learning disabilities.

    Cases will be purposively chosen to include key sub-groups of the wider population of autistic people and people with learning disabilities. The sample will be inclusive of (1) children and adults, (2) autistic children and adults, and children and adults with learning disabilities including those with mild, moderate and severe learning disabilities, and (3) those from specialist assessment and treatment inpatient services, forensic services, and generic inpatient mental health services for both children and adults. Data on protected characteristics including disability, sex, and ethnicity will be collected. The investigators will make use of translators and translation as needed, and an associated budget has been included.

    Stage 3 (Work Package 4) Anonymous data about autistic inpatients and inpatients with learning disabilities from (i) Assuring Transformation, and (ii) Mental Health Services datasets. These data are freely available from NHS Digital and are fully anonymised.

    Stage 4 (Work Package 5) This final stage will make use of data drawn from all aforementioned Stages.

    Identification of Services and Participants

    Stage 1 (Work Package 1) NHS Trusts, social care providers, private sector hospitals and services in England providing mental health and learning disabilities services to those with autism and/or learning disabilities will be eligible for inclusion.

    Participants will be approached via posters, social media postings, emails, and text messages. Such information about how to take part will be disseminated through Integrated Care Boards, Provider Collaboratives, commissioners, NHS Trusts, local authorities, and social care providers nationally, including inpatient services and community teams. Further information about the survey will be shared by the National Autistic Society, Challenging Behaviour Foundation, and Learning Disability England directly with and through networks of carers, family members, and people with learning disabilities, and autistic people. Younger child participants will be identified via an item in the parent/carer survey asking if they would be comfortable being contacted about potential data collection from the child who has received a C(E)TR that they are completing the survey about - with various options of how such data collection can occur to meet the individual communication needs of the child (including full survey, shorter version of the survey, or Talking Mats® interview).

    Stage 1 (Work Package 2) Participants will be approached via posters, social media postings, emails, and text messages. Such information about how to take part will be disseminated through Integrated Care Boards, Provider Collaboratives, commissioners, NHS Trusts, local authorities, and social care providers nationally, including inpatient services and community teams and NHS England. The survey will also be promoted by the National Autistic Society, Challenging Behaviour Foundation, and Learning Disability England including through relevant professional networks.

    Stage 2 (Work Package 3) NHS Trusts and private sector hospitals in England providing inpatient psychiatric care to autistic people and people with learning disabilities will be eligible for inclusion.

    The investigators will disseminate information about the study to Integrated Care Boards, Provider Collaboratives, private sector hospitals, commissioners, NHS Trusts, local authorities and social care providers nationally. Study research will also be promoted by the National Autistic Society, Challenging Behaviour Foundation, and Learning Disability England to help ensure maximum reach. The investigators will then work directly with services that express interest to identify potential cases.

    Stage 3 (Work Package 4) Anonymous data from (i) Assuring Transformation, and (ii) Mental Health Services datasets will be accessed. These data are freely available for download from NHS Digital and currently within the public domain.

    Stage 4 (Work Package 5) N/A

    Study procedures

    Stage 1 (Work Package 1) Potential survey participants will have been approached with research information. Potential participants will have been provided with an information sheet about the study, with which to decide about whether they would like to take part in the research. They will also be encouraged to contact the research team if they have any additional questions or would like any further information to make an informed decision of whether to take part in the research. Interested participants will be given options of how they would prefer to complete the survey, including independently online or receiving support to complete the survey. Options for support include: (i) text to speech reader, (ii) easier-to-read text, (iii) having someone present to provide support, (iv) manual sign support and (v) translation into languages other than English.

    When expressing a preference about how to complete the survey, participants will provide identifiable contact details. These will include their name, and contact details including postal address, email address, and phone number as per their preference of how they would like us to contact them. The primary rationale for the surveys not being anonymous is to guard against fraudulent responses (e.g., ineligible people completing the survey purely to receive the voucher). By having a small amount of contact with participants between them expressing interest and completing the survey there is a greater chance of identifying fraudulent responses. A secondary rationale is that the investigators need identifiable personal data to fulfil duty of care and safeguarding obligations (e.g., if a disclosure was made within a survey, the investigators would not be able to act on this if they did not know personal information). Additionally, to send participant vouchers, the investigators need to know their name and address.

    Potential child participants will have been identified via an item in the parent/carer survey asking if they would be comfortable being contacted about potential data collection from the child who has received a C(E)TR that they are completing the survey about. It would then be discussed with the parent/carer what would be the most suitable format for the child to provide data - including completing the full survey, a shorter version of the survey, or a Talking Mats® interview. The additional format options detailed above (e.g., text to speech reader, easier-to-read text, additional support from parent or carer) will also be considered. The focus will be on being guided by the family/child to adapt communication to meet the needs of the child, so that their voice can be included within the research.

    Having received expressions of interest the investigators will arrange for participants to complete the survey in accordance with their preferences (e.g., sending them a link to complete independently or providing desired support to complete the survey). Survey data will be captured on a single occasion where possible. The online surveys will be a blend of closed and open questions focused upon experiences of taking part within C(E)TRs, how they were carried out, the interface with dynamic support registers, perceived barriers and facilitators to participation, and the adjustments and supports made to support participation and empowerment along with any changes made to mental health services received. The investigators will make use of augmentative and alternative communication methods with younger children, and specifically, will complete Talking Mats® interviews. These will focus upon the experience of being admitted to hospital, if this occurred, and their experience of taking part in a C(E)TR, if they were included. The investigators recognise that younger children are unlikely to have been included within C(E)TRs, but they may have communicated their wishes; for example, they may have indicated that they wish to leave hospital and return home, and will aim to attempt to capture their voice about their experiences. The survey and interview questions will be further chosen and refined collaboratively with the LEAPs. For health economic analysis, questions to describe resources typically required to provide C(E)TRs and changes to the care pathway will also be asked.

    After completing the survey, participants will be shown a debrief sheet in the same manner that they have chosen to complete the survey e.g., text-to-speech reader, easier-to read text. This will detail their right to withdraw data and include a link to the online withdrawal form.

    Additional interviews with participants with moderate to severe learning disabilities will make use of augmentative and alternative communication methods to support the communication of participants as appropriate to their needs, such as Talking Mats® (www.talkingmats.com) and manual sign support (https://makaton.org) to aid processing and decision-making, including visually enhanced rating scales with optional tactile markers for those with no to limited vision. Before the visit some background information from participants and carers to generate a communication profile which can be used to support the interview will be collected.

    Talking Mats® uses questions that can be answered on a 3-point rating scale with picture symbols that are used to represent the topics, options, and the rating scale. Further, and to cater for the diverse communication needs of participants, the investigators will make use of the "easy on the i" image library which was developed by services for people with learning disabilities within Leeds and York Partnership NHS Foundation Trust and are available for use free of charge when using Talking Mats®. These pictures are coloured line drawings with text displayed above the image. The choice of image, topics, options, and ratings scales will be discussed and considered within the LEAPs. Each Talking Mat® is represented by a topic card, for example, "My Treatment" and a 3-point picture-based semantic rating scale is used representing good-ok-bad. Option cards associated with the topic are presented one by one to the participant who is invited to place each card within proximity to their preferred rating.

    Interviews will take place in the participant's setting. The Interviewer will sit at a table - ideally adjacent to the participant depending upon their needs. Talking Mat® symbol wallets will be placed to the outside of the interviewer to minimise distractions for the participant. The process is videoed with a video camera set up on tripod angled towards where the Talking Mat® will be carried out. The view should include both participant and interviewer as well as the Talking Mat® on the tabletop, and once completed, a digital photograph is taken of the completed Talking Mat®. An effectiveness rating tool is used across five domains to ensure that the participant's answers have been correctly understood [22]. The investigators are very experienced with the use of these methods within research.

    After consultee advice in the affirmative, Talking Mats® methodology will be used to determine assent/dissent from the person with moderate to severe learning disabilities (see Section 9.5). For those who confirm assent, the interview will then take place. Afterward, consultees will be shown a debrief sheet. This will detail their right to withdraw data and include a link to the online withdrawal form

    Stage 1 (Work Package 2) Potential survey participants will have been approached with research information Potential participants will have been provided with an information sheet about the study, with which to decide about whether they would like to take part in the research. They will also be encouraged to contact the research team if they have any additional questions or would like any further information to make an informed decision about whether to take part in the research. Interested participants will be given options of how they would prefer to complete the survey, including independently online or receiving support to complete the survey. Options for support include: (i) text to speech reader, (ii) easier-to-read text, (iii) having someone present to provide support, (iv) manual sign support , and (v) translation into languages other than English.

    When expressing a preference of how to complete the survey, participants will provide identifiable contact details. These will include their name, and contact details including postal address, email address, and phone number as per their preference of how they would like us to contact them. The primary rationale for the surveys not being anonymous is to guard against fraudulent responses e.g., ineligible people completing the survey purely to receive the voucher. By having a small amount of contact with participants between them expressing interest and completing the survey there is a greater chance of identifying fraudulent responses. A secondary rationale is that identifiable personal data is needed to fulfil a duty of care and safeguarding obligations e.g., if a disclosure was made within a survey, the investigators would not be able to act on this if personal information were not known. Additionally, to send participant vouchers, names and addresses need to be known.

    Having received expressions of interest the investigators will arrange for participants to complete the survey in accordance with their preferences (e.g., sending them a link to complete independently or providing desired support to complete the survey). Data will be captured on a single occasion. The online surveys will be a blend of closed and open questions focused upon experiences of taking part within C(E)TRs, how they were carried out, views regarding how the skill mix may relate to outcomes, how EbE are included and supported, perceived barriers and facilitators to participation, how C(E)TRs are integrated within existing methods and the adjustments and supports made to support participation and empowerment of people with learning disabilities and autistic people. For health economic analysis, questions to describe resources typically required to provide C(E)TRs and changes to the care pathway will also be included.

    After completing the survey, participants will be shown a debrief sheet in the same manner that they have chosen to complete the survey e.g., text-to-speech reader, easier-to read text. This will detail their right to withdraw data and include a link to the online withdrawal form.

    Stage 2 (Work Package 3)

    Potential cases will have been approached with research information. Multiple types of data about each case will be captured over time from a mixture of direct observation and recording of C(E)TR and CPA meetings, and interviews with those who attended these meetings. The following data will be captured:
    1. Information about the individual, including demographic data, and details of their hospital admission(s) and care team
    2. Audio/video recordings (where possible) and transcripts from multiple C(E)TRs, CPAs, and other patient meetings to track participant progress within their care pathway
    3. Semi-structured interviews with participants following each meeting. These will include C(E)TR panel chairs, clinical members, advocates, responsible clinicians, other health and social care staff, along with the individual and their family members or carers. As already described, adapted methods to provide inclusion, participation, and data capture (e.g., Talking Mats® with children and those with moderate to severe learning disabilities) will be used. Data will be captured, and interviews will be carried out to cover approximately 60 meetings (2 C(E)TRs, and a CPA meeting per individual). The researchers anticipate conducting up to 180 interviews in total across the 20 cases with individuals, carers and family members, C(E)TR panel members, and health and social care professionals
    4. Data extracted from a documentary review of C(E)TR paperwork including the completed Key Line of Enquiry document and associated workbooks for panel members, EbEs, and C(E)TR planners completed by individuals themselves, along with CPA paperwork and minutes and documents of other relevant patient meetings (e.g., MDT meetings, extraordinary patient meetings)

    At the end of Stage 2, approximately 15 months after initial case recruitment, participants will be shown a debrief form. This will detail their right to withdraw data and include a link to the online withdrawal form.

    Stage 3 (Work Package 4)

    Data from the publicly available anonymous Assuring Transformation and Mental Health Services datasets will be downloaded from NHS Digital.

    The monthly Assuring Transformation data set details the number of autistic inpatients and inpatients with learning disabilities over time published by NHS Digital from 2015 onwards. This anonymised national dataset reports the number of pre-admission and post-admission C(E)TRs completed each month, along with other data detailing information about an inpatient's care pathway (e.g., use of advocacy, type of inpatient service, planned discharge date, length of stay, family involvement in care, local authority involvement in care). The Assuring Transformation dataset reports data about the use of inpatient beds specifically commissioned for use by autistic people or people with a learning disability.

    Additional anonymised data about psychiatric bed utilisation by people with learning disabilities and autistic people is available from the Mental Health Services Data Set which is also published on a monthly basis by NHS Digital and will be downloaded and included. This data set is wider and includes information about the use of psychiatric beds by people with learning disabilities or autistic people that are not specifically commissioned for use by this population (e.g., autistic people or people with learning disabilities on a general psychiatric ward).

    Stage 4 (Work Package 5) Quantitative and qualitative data from the prior four work packages, inclusive of the investigators' estimate of resource implications, will be integrated using triangulation techniques. The researchers are experienced with these methods. The findings will be used to inform the context of good practice guidance for C(E)TRs, outlining best practice for maximising participation for people with learning disabilities and autistic people and their families/carers, as well as Experts by experiences how to implement C(E)TR outcomes effectively to maximise progression along care pathways, and guidance to overcome barriers. This analysis will also inform a final version of a logic model for C(E)TRs as a key project output.

ELIGIBILITY:
Eligibility criteria

Participants across all stages and work packages are eligible if they meet the following work package-specific inclusion criteria, and the work package-specific exclusion criteria do not apply. All queries about participant eligibility should be directed to the Study Manager.

Stage 1 (Work Package 1)

Inclusion criteria:

1. A person with a learning disability, or an autistic person, or a family member or carer of an autistic person or person with a learning disability
2. Having received or taken part in a C(E)TR within the last 12-months including blue-light C(E)TRs
3. Aged 5 or older (i.e. eligible to attend school at Key Stage one)
4. For those aged 16 years and older who lack capacity to make a decision about taking part in this research, advice indicating that they should be included from either a personal or nominate consultee
5. For those aged 15 and younger, consent from the person or organisation with parental responsibility

Exclusion criteria:

1. Only having received or taken part in Independently Chaired Care (Education) and Treatment Reviews (IC(E)TRs) within the last 12-months. IC(E)TRs are only for those held within long-term segregation and are out of scope
2. Aged younger than 5 years

Stage 1 (Work Package 2)

Inclusion criteria:

1. A C(E)TR chair, clinical member, or EbE or a health or social care professional, or commissioner
2. Who has taken part in a C(E)TR within the last 12-months including blue-light C(E)TRs.

Exclusion criteria:

1. Staff who have only taken part in Independently Chaired Care (Education) and Treatment Reviews (IC(E)TRs) within the last 12-months. IC(E)TRs are only for those held within long-term segregation and are out of scope

Stage 2 (Work Package 3)

Inclusion criteria:

People with learning disabilities or autistic people:

1. Who are due to have at least two C(E)TRs within 15-months
2. Aged 5 or older (i.e. eligible to attend school at Key Stage one)
3. For those aged 16 and older who lack capacity to make a decision about taking part in this research, advice indicating that they should be included from either a personal or nominate consultee
4. For those aged 5 years and older, but aged 15 years or younger, consent from the person or organisation with parental responsibility

C(E)TR panel members:

1. A chair, Expert by experience or clinical member who is due to attend a C(E)TR for a person with a learning disability or an autistic person who is taking part in this research project

Health and social care professions:

1. A health and social care profession who is due to attend a C(E)TR or CPA for a person with a learning disability or an autistic person who is taking part in this research project

Carers and family members:

1. A carer or family member who is due to attend a C(E)TR or CPA for someone with a learning disability or autism who is taking part in this research project

Exclusion criteria:

People with learning disabilities or autistic people:

1. Aged younger than 5 years.

Stage 3 (Work Package 4)

Inclusion criteria:

1. A person with a learning disability, or an autistic person, included within the Assuring Transformation and Mental Health Services datasets.

Exclusion criteria:

None.

Stage 4 (Work Package 5) N/A

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People with learning disabilities and autistic people, including children and young people, families and carers, C(E)TR panel members, and health and social care professionals including commissioners.
Sampling Method: Non-Probability Sample
Enrollment: 695 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Experiences of all stakeholders, including people with learning disabilities and autistic people and their families, when taking part in C(E)TRs | National surveys will be open for 8 months from their launch; data collection for case studies and associated semi-structed interviews will open for 15 months from the point of recruitment.
  Data will be gathered through national surveys; attendance at C(E)TRs, and CPA meetings to track individual progress over time, the collection of naturalistic data from the meetings, and though semi-structured interviews with attendees; and anonymised data available from NHS Digital for children and adults.

IPD SHARING:
Plan to Share IPD: No
The major output from this study will be the publication of good practice guidance for C(E)TRs developed in collaboration with our LEAPs and based upon our research findings inclusive of a logic model about the C(E)TR process. In accordance with our ethics approval the research team will act to preserve participant confidentiality and will not disclose or reproduce any information by which participants could be identified, except where specific consent is obtained, or if abusive practice is disclosed that researchers would have a duty to report. Individual participant data therefore will not be shared with other researchers. However, we will make a pseudonymised version of our data available following a reasonable request (i.e. not placed in the public domain).